CLINICAL TRIAL: NCT02977819
Title: Interventional Study in Cognitively Intact Seniors Aiming to Assess the Effects of Meditation Training and Foreign Language Learning on Behavioral, Biological and Neuroimaging Measures
Brief Title: Study in Cognitively Intact Seniors Aiming to Assess the Effects of Meditation Training
Acronym: Age-Well
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C16-38; 2016-A01767-44 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-11-04; First posted 2016-11-30 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meditation program (Experimental): Meditation courses and at-home practice
  Interventions: Other: Meditation practice
- English learning courses (Active Comparator): English learning courses and at-home practice
  Interventions: Other: Learning English as a foreign language
- No intervention (No Intervention): Follow-up without Meditation courses or English Learning courses

INTERVENTIONS:
Other: Meditation practice — 18 months
  Arms: Meditation program
Other: Learning English as a foreign language — 18 months
  Arms: English learning courses

SUMMARY:
As the number of older people in Europe grows, increasing healthy life years is a priority. As people live longer, ensuring good mental as well as physical health into later years is becoming ever more important. Cognitive decline, dementia (e.g. Alzheimer's Disease, AD), sleep disturbances and depression, all related to psychological distress and anxiety, are significant drivers of reduced quality of life in older adults. This project builds on evidence that meditation practice have the potential to downregulate these adverse factors and positively impact mental and neurological conditions including AD.

DETAILED DESCRIPTION:
Understanding of the neurocognitive mechanisms of meditation is still limited. Meditation can be conceptualized as "a set of complex emotional and attentional regulation strategies developed for a variety of purposes including the development of emotional well-being and balance". Affective (emotional) and cognitive (attentional) control are therefore the most likely mechanisms by which meditation could impact aging and AD. Specifically, meditation could enhance the controlling role of mid-brain structures and the executive network over structures involved in memory, emotions, and regulation of the immune system. This would lead to better emotional and cognitive control which in turn would be associated with improved mental and physical health.

ELIGIBILITY:
1. Inclusion Criteria :

   For all participants
   * Age ≥ 65 years ;
   * To be autonomous
   * Live in their home;
   * Educational level ≥ 7 years (from the Preparatory Course (First grade) included);
   * To be registered to the social security system ;
   * To be motivated to effectively participate in the project and to sign the consent form in agreement with the local ethic committee ;
   * Neuropsychological performances within the normal range (according to age, sex, and educational level), as assessed by the diagnostic battery.

   For participants without previous meditation practice
   * French mother tongue;
   * Available for the trial duration (24 months);
   * Retired since 1 year or more;
   * No preference regarding the intervention group ;
   * Not having regularly or intensively practiced meditation or comparable practices (yoga, Qi Gong, Alexander technique) as follows :

     * more than one day per week for more than six months consecutively over the last 10 years,
     * intensively (internship or retreat > five consecutive days) over the past 10 years,
     * more than 25 days of retreats (cumulatively) prior to the last 10 years ;
   * Not speaking English fluently.

   For expert meditators :
   * Formal meditation practice > 10 000 hours in the whole life, including at least 6 cumulated months of retreat;
   * Daily meditation practice (at least 6 days/week, 45 minutes/day);
   * Mindfulness meditation practice (i.e. mindfulness, samatha/vipassana, zazen (zen), shikantaza (zen), focused attention, mahamudra/Dzogchen, and compassion/loving jindness (tonglen, metta/karuna, bodhichitta)
2. Exclusion criteria :

   * Contraindication to MRI or PET Amyvid® ;
   * For security reasons realted with the use of Amyvid®, a blood sampling allowing to measure hepatic and renal functions will be performed at the V1 visit before the PET-Amyvid® scan. In case anomalies are detected of grade 3 or higher severity, the PET-Amyvid® scan will not be performed.
   * Hypersensitivity to Amyvid®
   * History or presence of a major neurological or psychiatric disorder (including an addiction to alcohol or drugs);
   * History of cerebral disease (vascular, degenerative, physical malformation, tumor, or head trauma with loss of consciousness for more than an hour);
   * Presence of a chronic disease or acute unstable illness (respiratory, cardiovascular, digestive, renal, metabolic, hematologic, endocrine or infectious);
   * Current or recent medication that may interfere with cognitive action or radiological measures (psychotropic drugs, antihistamines, anti-Parkinsonian drugs, benzodiazepines, non-steroidal anti-inflammatory agents, antiepileptics, central analgesic and muscle relaxants);
   * Under legal guardianship or incapacitation;
   * Inclusion in another biomedical research protocol at baseline, if including use of a radiolabel for radiological measures;
   * Physical of behavioural inhabilities to perform the follow-up visits as planned in the study protocol.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Estimate the effect of an 18-month meditation intervention in non-meditating senior participants on the volume of the anterior cingulate cortex compared to a passive control intervention | Visit 1 inclusion - Visit 3 Month 18
  change in anterior cingulate cortex volume (T1-weighted MRI)
Estimate the effect of an 18-month meditation intervention in non-meditating senior participants on the perfusion of the anterior cingulate cortex compared to a passive control intervention | Visit 1 inclusion - Visit 3 Month 18
  change in anterior cingulate cortex perfusion (early PET-Amyvid® scan)
Estimate the effect of an 18-month meditation intervention in non-meditating seniors on the volume of the insula compared to an 18 months intervention of learning a foreign language | Visit 1 inclusion - Visit 3 Month 18
  change in insula volume (T1-weighted MRI)
Estimate the effect of an 18-month meditation intervention in non-meditating seniors on the perfusion of the insula compared to an 18 months intervention of learning a foreign language | Visit 1 inclusion - Visit 3 Month 18
  change in insula perfusion (early PET-Amyvid® scan)

SECONDARY OUTCOMES:
Comparison between meditation intervention and language learning intervention on the global metacognitive composite score | up to 35 months post intervention
  consisting in the mean of the attentional, constructive and deconstructive subscores (main behavioural outcome) Each composite score is computed by averaging its respective standardised scale scores (range (-3) - (4) , Higher score of the meditation composite score mean better outcome)
Composite score per cognitive area assessed by the neuropsychological tests and the questionnaires | up to 35 months post intervention
  composite scores will be computed as z-scores calculated from all the cognitive scores obtained for the corresponding cognitive function that will have a normal distribution and will not have a floor or ceiling effect. Additional exploratory analyses will be conducted on all individual behavioural measures obtained.
Medical neuroimaging using MRI: grey and white matter volume in all brain voxels | up to 35 months post intervention
  grey and white matter volume in all brain voxels
Medical neuroimaging using MRI: hippocampal and hippocampal subfield volumes | up to 35 months post intervention
  hippocampal and hippocampal subfield volumes
Medical neuroimaging using MRI: brain perfusion in all brain voxels | up to 35 months post intervention
  brain perfusion in all brain voxels
Medical neuroimaging using MRI: fractional anisotropy and mean diffusivity in all brain voxels | up to 35 months post intervention
  fractional anisotropy and mean diffusivity in all brain voxels
Medical neuroimaging using MRI: number, size, type and location of white matter lesions | up to 35 months post intervention
  number, size, type and location of white matter lesions
Medical neuroimaging using MRI: magnetic susceptibility index in all brain voxels | up to 35 months post intervention
  magnetic susceptibility index in all brain voxels
Medical neuroimaging using MRI: brain functional connectivity measures in all brain voxels at rest in a non-meditative state | up to 35 months post intervention
  brain functional connectivity measures in all brain voxels at rest in a non-meditative state
Beta-amyloid charge (of the radiopharmarceutical Amyvid®) measured in each voxel of the brain and gross mean in gray matter | up to 35 months post intervention
  measured in each voxel of the brain and gross mean in gray matter
Glucose Cerebral Consumption at rest (relative to mean consumption measured in the cerebellum) | up to 35 months post intervention
  Glucose Cerebral Consumption at rest (relative to mean consumption measured in the cerebellum) by TEP
Medical neuroimaging using fMRI: Brain activity specifically associated with emotional processes (comparing emotional to neutral items) during the Rest-SoVT task. | up to 35 months post intervention
  Brain activity specifically associated with emotional processes (comparing emotional to neutral items) during the Rest-SoVT task.
Medical neuroimaging using fMRI: Brain activity specifically associated with attentional processes (altertness, inhibition, sustained attention) during the AX-CPT task. | up to 35 months post intervention
  Brain activity specifically associated with attentional processes (altertness, inhibition, sustained attention) during the AX-CPT task.
Medical neuroimaging using PET-scan and Amyvid® radiotracer | up to 35 months post intervention
  Brain amyloid load (of the PET-Amyvid® radiotracer) measured in global grey matter mask
Subjectives sleep measures with sleep quality index z-score mean of the scores at questionnaires | up to 35 months post intervention
  Epworth scale, Leeds Sleep evaluation questionnaire, Pittsburg Sleep Quality Scale, St Mary's hospital questionnaire, Berlin Questionnaire, and Insomnia severity index.
Mean duration of sleep | up to 35 months post intervention
  Data collected by actimetrics record
fragmentation indices during activity and resting states | up to 35 months post intervention
  Data collected by actimetrics record
regularity of the rest-activity cycle | up to 35 months post intervention
  Data collected by actimetrics record
Mean z-score of total sleep time | up to 35 months post intervention
  Data collected during polysomnographic sleep record with Somno-Art device
Mean z-score of sleep onset latency | up to 35 months post intervention
  Data collected during polysomnographic sleep record with Somno-Art device
Mean z-score of sleep efficiency | up to 35 months post intervention
  Data collected during polysomnographic sleep record with Somno-Art device
Biological blood tests | up to 35 months post intervention
  tau, phosphotau, Ab 40, 42, APOE4, NFL, BDNF, GWAS, cytokines, CRP, cortisol, serotonine, SDHEA, SHBG, E2, testosterone, glycemie, insuline, BNP, tPA, PAI-1, peroxyredoxine
Telomerase properties by blood tests | visit 1 baseline -Visit 3 18 months
  Telomerasic activity, telomerase length
lymphocytic immunophenotyping | visit 1 baseline -Visit 3 18 months
  biological blood tests
Difference in partner perceptions of participant mindfulness measured by Five-Facet Mindfulness Questionnaire (FFMQ-15, range 15-75, higher scores indicate greater mindfulness) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant.
Difference in partner perceptions of participant compassion towards others measured by Compassionate Love Scale (Range 21-147, higher scores indicate greater compassion) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant
Difference in partner perceptions of participant depression measured by the Geriatric Depression Scale (range 0-15, higher scores indicate greater depressive symptoms) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant
Scores to evaluate the impact on volunteers' relatives | up to 35 months post intervention
  scores to hetero questionnaires fulfilled by relatives and qualitative data from interviews with the participants on one hand and with the teachers on the other hand
Difference in partner perceptions of participant anxiety measured by trait subscale of the state-trait anxiety inventory (trait-STAI, range 20-80, higher scores indicate greater anxiety symptoms) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant
Difference in partner perceptions of participant prosocialness measured by Prosocialness scale (range 16-80, higher scores indicate greater prosocialness) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant
Difference in partner perceptions of participant's cognitive difficulties in everyday life, measured by Mc Nair CDS (range 0-156, higher score indicates greater cognitive difficulties) | up to 35 months post intervention
  Partners are defined as spouse, sibling, child, neighbour or friend in close contact with the participant
Neural signature of meditative practices using brain medical imaging (neuronal activity in each cerebral voxel (fMRI) at rest and during the emotional task, in a mindfulness meditative state versus not; in compasional meditative state or not) | up to 35 months post intervention
  only for meditation experts
Safety and acceptance | up to 35 months post intervention
  recording adverse events, measurement of anxiety, depression, satisfaction, and well-being using questionnaires
evaluation of the practice of the meditation practice and language learning at long-term (29 months post-intervention) | up to 35 months post intervention (because V4 = 29 months post intervention with a window of 6 months
  questionnaire about the practice (meditation or foreign language)
Behavioral measures (questionnaires) to evaluate the psychological impact of the confinement | up to 35 months post intervention
  composite score per function (anxiety, stress, auto-compassion...)

CONTACTS AND LOCATIONS:
Overall Officials: De La Sayette Vincent, Principal Investigator — CHU Caen - France; Chételat Gaël, Study Director — GIP Cyceron Caen
Locations (1):
- GIP Cyceron, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: Yes
Data access of AGE-WELL and SCD-WELL studies of the MEDIT-AGEING project for which Institut national de la santé et de la recherche médicale (Inserm) is the sponsor. The Material can be mobilized, under the conditions and modalities defined in the Charter, by any research team belonging to an Academic signatory to the Consortium Agreement concluded for the needs of the Project or by any research team belonging to an Academic outside the Consortium Agreement, French or foreign, for carrying out SRP relating to the scientific theme of mental health and wellbeing in older people.
  The Material may also be mobilized, by non-academic third parties for the realization of SRP relating to the scientific theme of mental health and wellbeing in older people, under conditions, in particular financial, which will be established by separate agreement between Inserm and by the said third party.
Supporting Information: Study Protocol
Time Frame: December 2020
Access Criteria: * specific information (quantity of Data available on a given date, number of patients included in the Cohort meeting the specific selection criteria for SRP requests, etc.) necessary for the conception of the SRP request;
  * the price list for the mobilization of Data within the framework of the SRP.
  * the list of services likely to be performed by the signatories of the Consortium Agreement for the purposes of the SRP request, as well as the associated price list;
  * a quote for services not included in the price list.
URL: https://silversantestudy.fr/

REFERENCES:
- [Background] Chetelat G, Lutz A, Klimecki O, Frison E, Asselineau J, Schlosser M, Arenaza-Urquijo EM, Mezenge F, Kuhn E, Moulinet I, Touron E, Dautricourt S, Andre C, Palix C, Ourry V, Felisatti F, Gonneaud J, Landeau B, Rauchs G, Chocat A, Quillard A, Devouge EF, Vuilleumier P, de La Sayette V, Vivien D, Collette F, Poisnel G, Marchant NL; Medit-Ageing Research Group. Effect of an 18-Month Meditation Training on Regional Brain Volume and Perfusion in Older Adults: The Age-Well Randomized Clinical Trial. JAMA Neurol. 2022 Nov 1;79(11):1165-1174. doi: 10.1001/jamaneurol.2022.3185. PMID 36215061
- [Background] Schlosser M, Klimecki OM, Collette F, Gonneaud J, Kliegel M, Marchant NL, Chetelat G, Lutz A; Medit-Ageing Research Group. An 18-month meditation training selectively improves psychological well-being in older adults: A secondary analysis of a randomised controlled trial. PLoS One. 2023 Dec 1;18(12):e0294753. doi: 10.1371/journal.pone.0294753. eCollection 2023. PMID 38039341
- [Background] Poisnel G, Arenaza-Urquijo E, Collette F, Klimecki OM, Marchant NL, Wirth M, de La Sayette V, Rauchs G, Salmon E, Vuilleumier P, Frison E, Maillard A, Vivien D, Lutz A, Chetelat G; Medit-Ageing Research Group. The Age-Well randomized controlled trial of the Medit-Ageing European project: Effect of meditation or foreign language training on brain and mental health in older adults. Alzheimers Dement (N Y). 2018 Dec 14;4:714-723. doi: 10.1016/j.trci.2018.10.011. eCollection 2018. PMID 30581977
- [Derived] Haudry S, Dautricourt S, Gonneaud J, Landeau B, Calhoun VD, de Flores R, Poisnel G, Bougacha S, Kuhn E, Touron E, Chauveau L, Felisatti F, Palix C, Vivien D, de la Sayette V, Lutz A, Chetelat G. Effects of an 18-month meditation training on dynamic functional connectivity states in older adults: Secondary analyses from the Age-Well randomized controlled trial. Imaging Neurosci (Camb). 2025 Jun 10;3:IMAG.a.33. doi: 10.1162/IMAG.a.33. eCollection 2025. PMID 40800757
- [Derived] Champetier P, Hamel A, Andre C, Ourry V, Lacroix T, Rehel S, Chauveau L, Haudry S, Bertran F, de la Sayette V, Vivien D, Chetelat G, Lutz A, Rauchs G; Medit-Ageing Research Group. EEG Brain Rhythms During Resting-State Wakefulness and Sleep in Elderly Expert Meditators. J Sleep Res. 2025 Jul 29:e70161. doi: 10.1111/jsr.70161. Online ahead of print. PMID 40731281
- [Derived] Chauveau L, Gonneaud J, Poisnel G, Landeau B, Garnier-Crussard A, Pitel AL, Roquet D, Touron E, Haudry S, Mezenge F, Chocat A, Vivien D, de La Sayette V, Chetelat G, de Flores R; Medit-Ageing Research Group. Cardiovascular risk factors are associated with lower posterior-medial network functional connectivity in older adults. Alzheimers Res Ther. 2025 Jul 15;17(1):159. doi: 10.1186/s13195-025-01808-5. PMID 40665410
- [Derived] Requier F, Mohammadi H, Demnitz-King H, Schlosser M, Poisnel G, Salmon E, Chetelat G, Marchant NL, Lutz A, Collette F; Medit-Ageing Research Group. Examining cognitive differences in expert meditators and non-meditators older adults. Sci Rep. 2025 May 15;15(1):16898. doi: 10.1038/s41598-025-00226-9. PMID 40374672
- [Derived] Touron E, de Flores R, Coulbault L, Palix C, Chocat A, Kuhn E, Landeau B, Mezenge F, Roquet D, Chauveau L, Haudry S, Vivien D, de La Sayette V, Marchant NL, Chetelat G, Poisnel G; Medit-Ageing Research Group. Depressive symptoms in older adults are associated with changes in stress-related markers, functional connectivity and brain volume. Alzheimers Res Ther. 2025 Jan 6;17(1):9. doi: 10.1186/s13195-024-01643-0. PMID 39762947
- [Derived] Garnier-Crussard A, Gonneaud J, Felisatti F, Palix C, Ferrand Devouge E, Chocat A, Rauchs G, de la Sayette V, Vivien D, Demnitz-King H, Lutz A, Chetelat G, Poisnel G; Medit-Ageing Research Group. Effect of an 18-month meditation training on cardiovascular risk in older adults: a secondary analysis of the Age-Well randomized controlled trial. BMC Geriatr. 2024 Nov 16;24(1):954. doi: 10.1186/s12877-024-05550-9. PMID 39550530
- [Derived] Champetier P, Andre C, Rehel S, Ourry V, Landeau B, Mezenge F, Roquet D, Vivien D, de La Sayette V, Chetelat G, Rauchs G; Medit-Ageing Research Group. Multimodal neuroimaging correlates of spectral power in NREM sleep delta sub-bands in cognitively unimpaired older adults. Sleep. 2024 Apr 12;47(4):zsae012. doi: 10.1093/sleep/zsae012. PMID 38227830
- [Derived] Ourry V, Rehel S, Andre C, Mary A, Paly L, Delarue M, Requier F, Hendy A, Collette F, Marchant NL, Felisatti F, Palix C, Vivien D, de la Sayette V, Chetelat G, Gonneaud J, Rauchs G; Medit-Ageing Research Group. Effect of cognitive reserve on the association between slow wave sleep and cognition in community-dwelling older adults. Aging (Albany NY). 2023 Sep 28;15(18):9275-9292. doi: 10.18632/aging.204943. Epub 2023 Sep 28. PMID 37770186
- [Derived] Demnitz-King H, Requier F, Whitfield T, Schlosser M, Gonneaud J, Ware C, Barnhofer T, Coll-Padros N, Dautricourt S, Delarue M, Klimecki OM, Paly L, Salmon E, Schild AK, Wirth M, Frison E, Lutz A, Chetelat G, Collette F, Marchant NL; Medit-Ageing Research Group. Effects of Meditation Training and Non-Native Language Training on Cognition in Older Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2317848. doi: 10.1001/jamanetworkopen.2023.17848. PMID 37450303
- [Derived] Andre C, Kuhn E, Rehel S, Ourry V, Demeilliez-Servouin S, Palix C, Felisatti F, Champetier P, Dautricourt S, Yushkevich P, Vivien D, de La Sayette V, Chetelat G, de Flores R, Rauchs G; Medit-Ageing Research Group. Association of Sleep-Disordered Breathing and Medial Temporal Lobe Atrophy in Cognitively Unimpaired Amyloid-Positive Older Adults. Neurology. 2023 Jul 25;101(4):e370-e385. doi: 10.1212/WNL.0000000000207421. Epub 2023 May 31. PMID 37258299
- [Derived] Champetier P, Andre C, Weber FD, Rehel S, Ourry V, Laniepce A, Lutz A, Bertran F, Cabe N, Pitel AL, Poisnel G, de la Sayette V, Vivien D, Chetelat G, Rauchs G. Age-related changes in fast spindle clustering during non-rapid eye movement sleep and their relevance for memory consolidation. Sleep. 2023 May 10;46(5):zsac282. doi: 10.1093/sleep/zsac282. PMID 36433753
- [Derived] Demnitz-King H, Gonneaud J, Klimecki OM, Chocat A, Collette F, Dautricourt S, Jessen F, Krolak-Salmon P, Lutz A, Morse RM, Molinuevo JL, Poisnel G, Touron E, Wirth M, Walker Z, Chetelat G, Marchant NL; Medit-Ageing Research Group. Association of Self-reflection With Cognition and Brain Health in Cognitively Unimpaired Older Adults. Neurology. 2022 Sep 27;99(13):e1422-e1431. doi: 10.1212/WNL.0000000000200951. Epub 2022 Jul 19. PMID 35853750
- [Derived] Felisatti F, Gonneaud J, Palix C, Garnier-Crussard A, Mezenge F, Landeau B, Chocat A, Quillard A, Ferrand-Devouge E, de La Sayette V, Vivien D, Chetelat G, Poisnel G; Medit-Ageing Research Group. Role of Cardiovascular Risk Factors on the Association Between Physical Activity and Brain Integrity Markers in Older Adults. Neurology. 2022 May 17;98(20):e2023-e2035. doi: 10.1212/WNL.0000000000200270. Epub 2022 Apr 13. PMID 35418459
- [Derived] Andre C, Rehel S, Kuhn E, Landeau B, Moulinet I, Touron E, Ourry V, Le Du G, Mezenge F, Tomadesso C, de Flores R, Bejanin A, Sherif S, Delcroix N, Manrique A, Abbas A, Marchant NL, Lutz A, Klimecki OM, Collette F, Arenaza-Urquijo EM, Poisnel G, Vivien D, Bertran F, de la Sayette V, Chetelat G, Rauchs G; Medit-Ageing Research Group. Association of Sleep-Disordered Breathing With Alzheimer Disease Biomarkers in Community-Dwelling Older Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2020 Jun 1;77(6):716-724. doi: 10.1001/jamaneurol.2020.0311. PMID 32202593